CLINICAL TRIAL: NCT06989606
Title: Burnout in UK Paramedics: a National Survey
Acronym: BURNS
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Jonathan Robinson, Ph.D, Senior Lecturer in Research Methods, Teesside University
Other Study IDs: 12818
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Burnout; Sleep; Paramedical Professional; Shift Work
Keywords: Burnout; Sleep Quality; Paramedic
MeSH Terms: conditions — Burnout, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to learn how common burnout is among UK paramedics and what factors are associated with it. It also aims to explore how burnout relates to sleep quality and the intention to leave the profession. The main questions it aims to answer are:

1. What is the prevalence of burnout among UK paramedics?
2. How is burnout related to sleep quality?
3. What personal or job-related factors are linked to higher levels of burnout?
4. Does burnout relate to paramedics' intentions to leave the profession?

Participants completed an online survey that included:

1. Demographic questions (e.g. age, years of service, shift patterns)
2. The Copenhagen Burnout Inventory (CBI) to assess burnout
3. The Pittsburgh Sleep Quality Index (PSQI) to measure sleep quality

Questions about their intention to leave the profession

Researchers analysed the responses using statistical techniques to identify relationships between burnout, sleep quality, and work-related factors.

DETAILED DESCRIPTION:
This cross-sectional observational study investigated the prevalence and associated factors of burnout among UK paramedics, with a particular focus on the relationship between burnout and sleep quality. The impetus for this research stems from increasing concerns about workforce sustainability within UK ambulance services, where high attrition rates and recruitment challenges have raised concerns about the occupational wellbeing of paramedics. Burnout and poor sleep quality are known to negatively impact both individual health and job performance, making this an urgent area for empirical study.

Data were collected via an anonymous online survey disseminated through the College of Paramedics and social media channels. The survey comprised demographic questions (e.g. age, gender, years of service, shift length, and number of calls attended), the Copenhagen Burnout Inventory (CBI) to assess personal, work-related, and client-related burnout, and the Pittsburgh Sleep Quality Index (PSQI) to evaluate various dimensions of sleep quality. The survey also included an item assessing intention to leave the profession.

There are approximately 22,000 registrants (full, student and associate members) to the CoP (CoP, 2021), representing the total potential sample size eligible to complete the survey. A power analysis using an online sample size calculator (http://www.raosoft.com/samplesize.html) - based on a 50% response distribution, a 5% margin of error, and an 80% confidence level - indicates that the required sample size will be 164. To adjust for incomplete data, the sample size has been increased by 10%, indicating a sample of 181.

Analyses were conducted using JASP. Descriptive statistics were used to summarise participant characteristics and prevalence rates. Correlational analyses (both frequentist and Bayesian) examined associations between burnout scores, sleep quality, and key demographic and occupational variables. Logistic regression was employed to explore predictors of burnout, including PSQI scores, shift duration, call volume, and years of service.

This study provides novel insights into the occupational wellbeing of UK paramedics, with implications for workforce planning, health promotion, and retention strategies within emergency medical services.

ELIGIBILITY:
Inclusion Criteria:

* A member of the College of Paramedics, and/or a qualified or student Paramedic.
* At least 18 years of age to be able to provide consent to take part in the online survey.
* Able to read and write in the English language.

Exclusion Criteria:

* Under the age of 18 years.
* Not a Paramedic (As associate members of the College of Paramedics are not required to be a paramedic).
* Not able to read and write in the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A member of the College of Paramedics, and/or a qualified or student Paramedic.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Copenhagen Burnout Inventory (CBI) questionnaire (Kristensen et al., 2005) | This was completed at a single time point, depending on when the voluntary participant completed the questionnaire (between 10 March 2023 and 21 April 2023).
  The CBI assesses three dimensions: personal burnout, work-related burnout, and client-related burnout. A contributing factor of burnout is sleeping pattern and quality. The PSQI assesses sleep quality and disturbances through seven subscales: sleep latency, sleep duration, sleep quality, sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. These seven domains of sleep quality can be summed to obtain a maximum achievable score of 21, which indicates the highest level of sleep disturbance.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) questionnaire (Buysse et al., 1989). | This was completed at a single time point, depending on when the voluntary participant completed the questionnaire (between 10 March 2023 and 21 April 2023).
  The PSQI assesses sleep quality and disturbances through seven subscales: sleep latency, sleep duration, sleep quality, sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. These seven domains of sleep quality can be summed to obtain a maximum achievable score of 21, which indicates the highest level of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Robinson, PhD, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No